CLINICAL TRIAL: NCT05109858
Title: Observational Study on Skin Toxicity by Oncological Therapies
Brief Title: Skin Toxicity by Oncological Therapies
Acronym: SKINTOX
Status: Completed | Type: Observational
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IRST100.41
Record Dates: First submitted 2021-09-16; First posted 2021-11-05 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Skin Toxicity
Keywords: skin toxicities; oncological therapies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter, retrospective and prospective observational study. The project involves the collection of clinical data of patients treated with oncological therapies, to evaluate skin toxicities related to oncological treatment.

DETAILED DESCRIPTION:
This is a multicenter, retrospective and prospective observational study. The research will include 300 patients treated with clinical practice oncological treatments (approved by Italian Competent Authority, AIFA) from January 2012 to February 2024.

Patients will follow the prescribed therapeutic indications according to regular clinical practice and data from their medical records will be collected in a study database.

Primary objective of the study is the evaluation of the type, frequency and severity of skin toxicities related to oncological treatment.

Secondary objectives are:

* Evaluation of the association between skin toxicities due to oncological treatment and drug activity and effectiveness parameters(ORR, PFS, OS);
* Evaluation of the association between clinical-pathological features of primary cancer and skin toxicities of oncological treatment;
* Evaluation of the optimal management of skin toxicities related to cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who have signed informed consent.
2. Consecutive retrospective patients and prospective patients treated with new clinical practice oncological treatments (approved by AIFA) from January 2012 to February 2024
3. Male or female, age ≥18 years.

Exclusion Criteria:

Participation in another clinical trial with any investigational drug.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with any oncological therapy (approved by AIFA) as per clinical practice, from 2012 to 2024.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of the type of skin toxicities related to oncological treatment | 5 years
  Data will be described using absolute and (percentage) relative frequencies calculated for specific types of skin toxicities collected by the participating centers. Specific types of skin toxicities will be defined during dermatologists involved in the study, based on subjects enrolled at each site.
Evaluation of the frequency of skin toxicities related to oncological treatment | 5 years
  Absolute and (percentage) relative frequencies will be calculated for skin toxicities, stratified considering different oncological treatments.
Evaluation of the severity of skin toxicities related to oncological treatment | 5 years
  Grade of severity of skin toxicities will be collected: absolute and (percentage) relative frequencies will be calculated for different grades of severity.

SECONDARY OUTCOMES:
Evaluation of the association between skin toxicities and baseline clinical parameters | 5 years
  A statistical model will be carried out, namely a mathematical relationship between presence of skin toxicities and baseline clinical parameter. Mathematical model will be a logistic regression, in which, independent variable is the presence of skin toxicities while dependent variables are parameters measured at baseline. These parameters could be continuous (for example: age of patients) or categorical (for example: gender or site of disease).
Evaluation of the association between skin toxicities and objective response rate | 5 years
  Statistical modelling of the association between skin toxicities and objective response rate (ORR) as drug effectiveness parameter. To analyze objective response rate (ORR), proportion of patients with complete and partial response will be calculated, globally for all patients and considering different subgroup of treatment type.
Evaluation of the association between skin toxicities and progression-free survival | 5 years
  Statistical modelling of the association between skin toxicities and progression-free survival (PFS) as drug effectiveness parameter. To evaluate progression-free survival, difference between date of start therapy and date of disease progression (or death) will be calculated.
Evaluation of the association between skin toxicities and overall survival | 5 years
  Statistical modelling of the association between skin toxicities and overall survival (OS) as drug effectiveness parameter. To evaluate overall survival, difference between date of start therapy and date of or death will be calculated. Time for patients without event (progression of disease or death) will be considered from date of start therapy and date of last contact.
Evaluation of the optimal management of skin toxicities related to cancer treatment | 5 years
  Data related to management of skin toxicities will be described using absolute and (percentage) relative frequencies calculated for specific types of skin toxicities collected by the participating centers.

CONTACTS AND LOCATIONS:
Overall Officials: Matelda Medri, PhD, Study Chair — IRST IRCCS
Locations (20):
- Italy (20):
  - Ospedale "Franz Tappeiner", Merano, Bolzano
  - AUSL della Romagna - Ospedale "M. Bufalini", Cesena, Forlì-Cesena
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST S.r.l., Meldola, Forlì-Cesena
  - Sapienza Università di Roma - Polo Pontino, Terracina, Latina
  - Centro di Riferimento Oncologico, Aviano, Pordenone
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari
  - IRCCS Istituto Tumori "Giovanni Paolo II", Bari
  - Università di Bologna, Bologna
  - Università "G. D'Annunzio", Chieti
  - Azienda USL Toscana Centro, Florence
  - ASL di Frosinone - Ospedale "Fabrizio Spaziani", Frosinone
  - Azienda Ospedaliera "Papardo", Messina
  - IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europe di Oncologia, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione "G. Pascale", Napoli
  - Università della Campania "Luigi Vanvitelli", Napoli
  - Università Campus Bio-Medico, Roma
  - Università degli Studi di Salerno AOU san Giovanni di Dio e Ruggi D'Aragona, Salerno
  - Azienda Ospedaliera Universitaria Senese, Siena
  - AOU Città della Salute e della Scienza, Torino